CLINICAL TRIAL: NCT06099392
Title: The Effect of Transcutaneous Electrical Acustimulation Combined With Polyethylene Glycol-electrolyte on the Quality of Small Bowel Preparation for Capsule Endoscopy
Brief Title: The Effect of Transcutaneous Electrical Acustimulation on Small Bowel Preparation for Capsule Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Wei-Fen Xie, Head of gastroenterology, Shanghai Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZXH202301
Record Dates: First submitted 2023-07-16; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Quality of Small Bowel Preparation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEA group (Experimental): TEA at ST36 (Zusanli) combined with 2L Polyethylene Glycol Electrolytes Powder for bowel preparation
  Interventions: Device: digital stimulators (SNM-FDC01, Ningbo MaidaMedical Device, Inc, Ningbo, China)
- Sham-TEA group (No Intervention): 2L Polyethylene Glycol Electrolytes Powder for bowel preparation

INTERVENTIONS:
Device: digital stimulators (SNM-FDC01, Ningbo MaidaMedical Device, Inc, Ningbo, China) — TEA at Zusanli(ST 36) 45 min when drinking Polyethylene Glycol Electrolytes Powder
  Arms: TEA group

SUMMARY:
Transcutaneous elctroacupuncture(TEA) at ST36 can improve gastrointestinal motility. Therefore,the investigators hypothesized that if TEA is applied to the preparation of small bowel capsule endoscopy, the small bowel peristalsis of patients can be regulated by electrical stimulation at (ST36). On the one hand, it can be used in combination with compound polyethylene glycol electrolyte powder, which is conducive to the discharge of small bowel contents and improve the imaging quality. On the other hand, it can improve the diagnostic rate by adjusting the intestinal transit time, And the completion rate of the examination can be improved by accelerating the gastric emptying time of capsule endoscopy.

Therefore, in order to explore the effect of TEA stimulation at ST36 combined with polyethylene glycol powder on preparation for small bowel capsule endoscopy, the investigators designed this study.

ELIGIBILITY:
Inclusion Criteria:

Agree to sign an informed consent form; Aged 18 to 75 years old Plan to undergo small bowel capsule endoscopy;

Exclusion Criteria:

Clinical diagnosis of gastrointestinal stricture, bowel obstruction, gastrointestinal fistula, intestinal resection; Clinical diagnosis of dysphagia; Those who require fasting or parenteral nutrition support treatment; Individuals with gastrointestinal motility disorders; Oral administration of gastrointestinal motility drugs within 1 week; Implanting medical electronic devices; Those who are allergic to compound polyethylene glycol electrolyte powder and dimethicone oil and cannot tolerate oral laxatives for intestinal preparation; Skin diseases that affect electrode fixation; Pregnant, preparing to conceive, or breastfeeding patients; Familiar with acupuncture and moxibustion treatment, acupoint selection or meridians; Researchers believe that it is not suitable for participants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
The rate of "adequate" cleansing of the small intestine | one year
  The rate of "adequate" cleansing of the small intestine

SECONDARY OUTCOMES:
Diagnostic rate of video capsule endoscopy | one year
  Diagnostic rate of video capsule endoscopy